CLINICAL TRIAL: NCT04334928
Title: Prevention of SARS-CoV-2 (COVID-19) Through Pre-Exposure Prophylaxis With Tenofovir Disoproxil Fumarate/Emtricitabine and Hydroxychloroquine in Healthcare Personnel: Randomized Clinical Trial Controlled With Placebo
Brief Title: Randomized Clinical Trial for the Prevention of SARS-CoV-2 Infection (COVID-19) in Healthcare Personnel
Acronym: EPICOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Plan Nacional sobre el Sida (PNS) (Other Government)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PrEP COVID-19
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Coronavirus Infection
Keywords: COVID-19; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomized double-blind clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Emtricitabine/Tenofovir (Experimental): Tenofovir Disoproxil Fumarate 245 mg/Emtricitabine 200 mg + Placebo of Hydroxychloroquine 200 mg
  1. Strength: 200 mg/245 mg tablets
  2. Dose: one tablet once a day (both at dinner)
  Interventions: Drug: Emtricitabine/tenofovir disoproxil; Drug: Placebo: Hydroxychloroquine
- Hydroxychloroquine (Experimental): Hydroxychloroquine 200 mg + Placebo of Tenofovir Disoproxil Fumarate 245 mg/Emtricitabine 200 mg
  1. Strength: 200 mg tablets
  2. Dose: one tablet once a day (both at dinner)
  Interventions: Drug: Hydroxychloroquine; Drug: Placebo: Emtricitabine/tenofovir disoproxil Placebo
- Emtricitabine/Tenofovir+Hydroxychloroquine (Experimental): Tenofovir Disoproxil Fumarate 245 mg/Emtricitabine 200 mg + Hydroxychloroquine 200 mg
  1. Strength FTC/TDF:200 mg/245 mg tablets
  2. Strength HC: 200 mg tablets
  3. Dose: one tablet FTC/TDF plus one tablet HC once a day (at dinner)
  Interventions: Drug: Emtricitabine/tenofovir disoproxil; Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Placebo of Tenofovir Disoproxil Fumarate 245 mg/Emtricitabine 200 mg + Placebo of Hydroxychloroquine 200 mg
  1. Placebo tablets with similar appearance to study drugs.
  2. Dose: one tablet once a day (both at dinner)
  Interventions: Drug: Placebo: Emtricitabine/tenofovir disoproxil Placebo; Drug: Placebo: Hydroxychloroquine

INTERVENTIONS:
Drug: Emtricitabine/tenofovir disoproxil — Emtricitabine/tenofovir disoproxil, 200 mg/245 mg tablets. A dose of one tablet once a day will be administered.
  Arms: Emtricitabine/Tenofovir; Emtricitabine/Tenofovir+Hydroxychloroquine
Drug: Hydroxychloroquine — Hydroxychloroquine, 200 mg tablets. A dose of one tablet once a day will be administered.
  Arms: Emtricitabine/Tenofovir+Hydroxychloroquine; Hydroxychloroquine
Drug: Placebo: Emtricitabine/tenofovir disoproxil Placebo — Placebo: Tablets similar in appearance to Emtricitabine/tenofovir disoproxil
  Arms: Hydroxychloroquine; Placebo
Drug: Placebo: Hydroxychloroquine — Placebo: Tablets similar in appearance to Hydroxychloroquine
  Arms: Emtricitabine/Tenofovir; Placebo

SUMMARY:
Healthcare workers are particularly at risk of SARS-CoV-2. This study aims to assess the efficacy of a daily single dose of tenofovir disoproxil fumarate (TDF) (245 mg)/ Emtricitabine (FTC) (200 mg), a daily single dose of hydroxychloroquine (HC) (200 mg), a daily single dose of TDF (245 mg)/FTC (200 mg) plus HC (200 mg) versus placebo, during 12 weeks in: (1) reducing the incidence of symptomatic disease and (2) reducing clinical severity COVID-19 among hospital healthcare workers aged 18 to 70 years in public and private hospitals in Spain.

DETAILED DESCRIPTION:
Healthcare workers are particularly at risk of SARS-CoV-2. In the absence of a vaccine, other strategies aiming to reduce the development of COVID-19 in the population, more specifically in healthcare workers is being sought. Administration of effective drugs to people at risk of developing an infectious disease is well accepted and is part of clinical practice. To date there are few on-going randomized clinical trial on Pre-exposure prophylaxis (PrEP) evaluating chloroquine and hydroxychloroquine efficacy for health care workers and other groups at high risk. Existing recent and scarce literature shows that RNA synthesis nucleos(t)ide analogue inhibitors, acting as viral RNA chain terminators, like TDF, abacavir or lamivudine, amongst others, could have an effect against SARS-CoV-2 infection. Worldwide, there is broad evidence of the use, safety and tolerability of hydroxychloroquine (200 mg) and TDF/FTC (245 mg/200 mg). This study aims to assess the efficacy of a daily single dose of TDF (245 mg)/FTC (200 mg), a daily single dose of HC (200 mg), a daily single dose of TDF (245 mg)/FTC (200 mg) plus HC (200 mg) versus placebo, during 12 weeks in: (1) reducing the incidence of symptomatic disease and (2) reducing clinical severity COVID-19 among hospital healthcare workers aged 18 to 70 years in public and private hospitals in Spain. Sample size calculations are based on the primary outcome; number of symptomatic confirmed infections by SARS-CoV-2. Briefly, 4.000 participants will be assigned to one of the 4 groups, through 1:1:1:1 randomization. Duration of prophylactic treatment will be 12 weeks from early April 2020 till early July 2020. Follow up of participants will continue up to 4 weeks after last dose of treatment. All participants will be assessed on a monthly basis. Interim analyses will be performed on monthly bases.

ELIGIBILITY:
Inclusion Criteria:

* Participants that, after receiving appropriate information on the study design, objectives, possible risks and acknowledging they have the right to withdraw from the study consent at any time, sing the informed consent for participation in the study.
* Male or female aged 18-70years.
* Health care workers in public or private hospitals in areas of risk of SARS-CoV-2 transmission.
* No previous diagnosis of SARS-CoV-2 (COVID-19) infection plus no symptoms compatible with SARS-CoV-2 (COVID-19) since 1st of March 2020 until the date of enrolment in the study.
* Understanding of the aim of the study and, therefore, acknowledging they have not been on any drug aiming at pre exposure prophylaxis against SARS-CoV-2 (COVID-19) since 1st of March 2020. This also includes PrEP for HIV.
* Negative pregnancy test during the previous 7 days to start treatments or more than 2 years after menopause.
* Women of reproductive age and their partners should commit to use and highly effective contraceptive method ( double barrier, hormonal contraception), during the study period and until 6 months after the last dose of treatment.

Exclusion Criteria:

* Having symptoms suggestive of COVID-19 infection
* HIV infection
* Active hepatitis B infection.
* Renal failure with estimated glomerular filtration rate (GFR) < 60 ml/min) and patients on Hemodialysis.
* Osteoporosis
* Myasthenia gravis
* Pre-existent maculopathy.
* Retinitis pigmentosa
* Bradycardia < 50bpm
* Weight < 40kg
* Participant with any immunosuppressive condition or hematological disease.
* Have taken any medications such as PrEP against SARS-CoV-2 from March 1, 2020 until trial entry (also includes PrEP for HIV).
* Treatment with drugs that may prolong QT in the last month before randomization for more than 7 days including: azithromycin, chlorpromazine, cisapride, clarithromycin, domperidone, droperidol, erythromycin, halofantrine, haloperidol, lumefantrine, mefloquine, methadone, pentamidine, procainamide, quinidine, quinine, sotalol, sparfloxacin, thioridazine, amiodarone.
* Breastfeeding
* Known allergy to any of the medication used in this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-07-11 (Actual)

PRIMARY OUTCOMES:
Number of confirmed symptomatic infections of SARS-CoV-2 (COVID-19) | 12 weeks

SECONDARY OUTCOMES:
Severity of disease in confirmed infected participants of SARS-CoV-2 (COVID-19) | 12 weeks
  assessed by:
  * No symptoms
  * Mild symptoms: general malaise, fever, cough, myalgia, asthenia.
  * Moderate symptoms: mild symptoms plus shortness of breath,
  * Severe symptoms: mild symptoms plus respiratory insufficiency that requires admission in intensive care unit and mechanical ventilation
Duration of symptoms in confirmed infected participants of SARS-CoV-2 (COVID-19) measured in days | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Polo, MD,PhD, Study Chair — Plan Nacional sobre el Sida (PNS); Miguel Hernán, MD,PhD, Study Chair — Harvard School of Public Health (HSPH)
Locations (65):
- Spain (65):
  - Hospital Universitario de Ferrol, Ferrol, A Coruña
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital General de Elche, Elche, Alicante
  - Hospital Sant Joan de Deu de Esplugues, Esplugues de Llobregat, Barcelona
  - Parc Sanitari Sant Joan de Déu de Sant Boi, Sant Boi de Llobregat, Barcelona
  - Hospital Moisès Broggi, Sant Joan Despí, Barcelona
  - Hospital Infanta Margarita, Cabra, Córdoba
  - Hospital Insular de Las Palmas, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Universitario de Canarias, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital de Donostia, San Sebastián, Guipuzcoa
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Fundación de Alcorcón, Alcorcón, Madrid
  - Hospital Colllado Villalba, Collado Villalba, Madrid
  - Hospital de Getafe, Getafe, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital de Móstoles, Móstoles, Madrid
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Hospital Quirón Pozuelo, Pozuelo de Alarcón, Madrid
  - Hospital de Torrejón, Torrejón de Ardoz, Madrid
  - Hospital Infanta Elena, Valdemoro, Madrid
  - Hospital Virgen del Castillo, Yecla, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Reina Sofía, Tudela, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Arnau de Vilanova, Llíria, Valencia
  - Hospital de Araba, Alava, Vitoria
  - Hospital General Universitario de Albacete, Albacete
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Centro Médico Teknon, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Dexeus, Barcelona
  - Hospital Quirón Barcelona, Barcelona
  - Hospital Universitario Sagrat Cor, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Virgen de la Luz, Cuenca
  - Hospital Clínico San Cecilio, Granada
  - Hospital Universitario de León, León
  - Hospital Universitario Ramón y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Reina Sofía, Murcia
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Complejo Asistencial de Palencia, Palencia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital General de Segovia, Segovia
  - Hospital Virgen del Rocio, Seville
  - Hospital Virgen Macarena, Seville
  - Hospital Clinico Universitario, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital General de Valencia, Valencia
  - Hospital La Fe, Valencia
  - Hospital de Valladolid, Valladolid
  - Hospital Rio Hortega, Valladolid
  - Hospital Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No